CLINICAL TRIAL: NCT02791568
Title: Advanced MRI for Uteroplacental Flow, Perfusion, Oxygenation & Inflammation
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-1222; A532800 (Other: UW Madison); SMPH\OBSTET & GYNECOL\OB-GYN (Other: UW Madison); 1U01HD087216-01 (NIH); Protocol Version 12/17/2019 (Other: UW Madison)
Record Dates: First submitted 2016-02-01; First posted 2016-06-07 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy; Obesity; Preeclampsia
MeSH Terms: conditions — Obesity; Pre-Eclampsia | interventions — High-Energy Shock Waves; Magnetic Resonance Spectroscopy; Ferrosoferric Oxide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pilot Study: 1. Ultrasound Scan
  2. MRI Scan
  3. Blood/Urine collection
  Interventions: Procedure: Ultrasound Scan; Procedure: MRI Scan
- Main Study- Control Group: 1. Ultrasound Scan
  2. MRI Scan
  3. Blood/Urine collection
  Interventions: Procedure: Ultrasound Scan; Procedure: MRI Scan
- Main Study- Study Group: 1. Ultrasound Scan
  2. MRI Scan
  3. Blood/Urine collection
  Interventions: Procedure: Ultrasound Scan; Procedure: MRI Scan
- Main Study- Ferumoxytol Group: 1. Ultrasound Scan
  2. MRI Scan
  3. Blood/Urine collection
  4. Ferumoxtyol Infusion
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Procedure: Ultrasound Scan — The research exam is expected to take 30 minutes for blood flow assessments
  Groups: Main Study- Control Group; Main Study- Study Group; Pilot Study
Procedure: MRI Scan — MR imaging will take approximately 30 minutes.
  Groups: Main Study- Control Group; Main Study- Study Group; Pilot Study
Drug: Ferumoxytol — A subset of subjects will complete MRI imaging with ferumoxytol as a contrast agent at the 24-28 week visit. A nurse will administer ferumoxytol in a hospital triage with pulse and blood pressure monitoring and fetal heart monitoring. The pharmacy will prepare the infusion and deliver to triage. Subjects will arrive at the obstetric triage unit for ferumoxytol injection three days prior to their scheduled ferumoxytol MRI study. In the triage, the nurse will obtain baseline vital signs and fetal heart rate. The IV Ferumoxytol infusion will be 30 minutes and atients will be monitored at 5 to 15-minute intervals. Three days after the ferumoxytol infusion, at 24-26 weeks gestation, subjects will have blood/urine collected, undergo a 30 minute ultrasound, a 30 minute MRI, an adverse event review, and medical record review. The MRI scanning procedure will be conducted at WIMR and will last approximately 30-60 minutes.
  Other Names: Feraheme®
  Groups: Main Study- Ferumoxytol Group

SUMMARY:
The purpose of the study is to develop advanced ultrasound (U/S) and Magnetic Resonance Imaging, known as MRI to study uteroplacental health. The goal of this study is to evaluate the blood and oxygen flow to the placenta using advanced U/S and MRI testing.

DETAILED DESCRIPTION:
Decreased uteroplacental perfusion is a recognized antecedent event in pregnancies that ultimately results in adverse outcomes like fetal growth restriction (FGR), preeclampsia (PE) and/or preterm birth. This concept is well supported clinically by identification of spiral artery vascular lesions called acute atherosis. Current literature suggests that these events occur very early which is why we are using multiple techniques related to flow at early time points. We are studying individuals with either poor maternal vascular response and/or inadequate spiral artery remodeling with resultant inadequate placentation will have a reduced uteroplacental perfusion. Given that the spiral arteries draw the vast majority of the blood flow in a gravid state, poor placentation would be reflected in the total uteroplacental blood flow (UPBF), and early detection would allow both design and then routine initiation of novel preventive therapies early in gestation to improve pregnancy outcome.

The goal of this research is to develop an arsenal of advanced ultrasound (U/S) and magnetic resonance imaging (MRI) techniques that are compatible to be run simultaneously or sequentially to probe uteroplacental health and overcome the limitations posed by obesity and motion. While safety concerns remain with MRI, particularly in the first trimester, we will front-load developmental and optimization studies in primate models as "proof of principle" before translating to humans; this conservative approach is key to our achieving paradigm shifting outcomes. A pilot study was completed prior to the main study to evaluate U/S Doppler and 2D PC MRI for UPBF measures that including contributions from the ovarian arteries in addition to the uterine arteries. The pilot study is now complete as the pilot data was evaluated after the enrolled pilot subjects completed the U/S and 2D PC MRI visits.

We are matching all imaging measures with clinical data and blood and urine sample post-hoc analyses for cytokines and tissue-specific metalloproteases, these correlations will further inform a differential diagnosis of distinct disease mechanisms that may otherwise show common imaging outcomes. At the end of the studies on both lean and obese women, we will inevitably have outcomes categorized as FGR, hypertensive and/or PE, perhaps preterm and/or rarely stillbirth outcomes. Using this combination of approaches we will determine: 1) an optimal combination of imaging methods that is practical and sufficiently safe to use in humans; 2) if new data so derived is informative beyond that currently available clinically; 3) at what point in gestation an abnormality may be detected by these new methods relative to current standard clinical measures and/or diagnoses; and 4) if imaging outcomes can predict specific complications, or only warn of a higher risk of general complications.

The primary objective of the ferumoxytol research, conducted under the pending Investigational New Drug Application, is to demonstrate homing of macrophages in vivo in the decidua of pregnancies with reduced uteroplacental blood-flow and perfusion. The secondary objective is to develop a test of placenta function in on-going pregnancies in subjects with reduced uteroplacental blood flow and perfusion. To evaluate these objectives, subjects with and without reduced total uterine blood-flow and possible reduced placental perfusion will receive Ferumoxytol (Feraheme®) prior to dynamic sequences magnetic resonance.

ELIGIBILITY:
Subject Population (Pilot study)

Inclusion Criteria:

1. Women with singleton, low-risk pregnancies
2. Gravida 1 (first pregnancy); or Gravida 2 (second pregnancy with first pregnancy carried to term or miscarried prior to 14 weeks or terminated); or Gravida 3 (third pregnancy with first and second pregnancies carried to term or one previous pregnancy carried to term and the other previous pregnancy miscarried prior to 14 weeks or terminated)
3. Ultrasound confirmed pregnancy dating prior to 14 weeks gestation
4. Non-obese (BMI 18.5-29.9 kg/M2) or Obese (Class I BMI 30-34.9 kg/M2 or Class II BMI 35-39.9 kg/M2) based on pregravid BMI

Exclusion Criteria:

1. Known fetal chromosome abnormality, structural malformation or syndromes in current pregnancy
2. Tobacco or alcohol or drug use in current pregnancy
3. Pre-existing autoimmune conditions or other maternal chronic diseases like renal diseases, chronic hypertension, thrombophilia, type I or II diabetes or any vasculopathy
4. History of sickle cell anemia or sickle cell trait
5. High risk for gestational hypertension, pre-eclampsia, HELLP syndrome, fetal growth restriction (FGR), abruptio placentae secondary to hypertension or pre-eclampsia, stillbirth/intrauterine fetal death

Subject Population (Main study) Inclusion Criteria

Control Group:

1. Non-obese (pregravid BMI 18.5-29.9 Kg/M2)25 (N=80)
2. Women with singleton, low-risk pregnancies
3. Gravida 1 (first pregnancy); or Gravida 2 (second pregnancy with first pregnancy carried to term or miscarried prior to 14 weeks or terminated); or Gravida 3 (third pregnancy with first and second pregnancies carried to term or one previous pregnancy carried to term and the other previous pregnancy miscarried prior to 14 weeks or terminated)
4. Ultrasound-confirmed pregnancy dating prior to 14 weeks gestation
5. Gestational age at screening prior to 16 weeks

Study Group:

1. Obese (pregravid Class I BMI 30-34.9 kg/M2 or pregravid Class II BMI 35-39.9 kg/M2) (N=80)
2. Women with singleton, low-risk pregnancies
3. Gravida 1 (first pregnancy); or Gravida 2 (second pregnancy with first pregnancy carried to term or miscarried prior to 14 weeks or terminated); or Gravida 3 (third pregnancy with first and second pregnancies carried to term or one previous pregnancy carried to term and the other previous pregnancy miscarried prior to 14 weeks or terminated)
4. Ultrasound confirmed pregnancy dating prior to 14 weeks gestation
5. Gestational age at screening prior to 16 weeks

Exclusion Criteria

Control and Study Groups:

1. Known fetal chromosome abnormality, structural malformation or syndromes in current pregnancy
2. Tobacco/alcohol/drug use in current pregnancy
3. Pre-existing autoimmune conditions or other maternal chronic diseases like renal diseases, chronic hypertension, thrombophilia, type I or II diabetes or any vasculopathy
4. History of sickle cell anemia or sickle cell trait
5. High risk for gestational hypertension, pre-eclampsia, HELLP syndrome, fetal growth restriction (FGR), abruptio placentae secondary to hypertension or pre-eclampsia, stillbirth/intrauterine fetal death

   a. The determination of whether or not the subjects are considered high risk for the conditions described above will be based on medical and obstetrical history review by clinical investigators with expertise in Maternal Fetal Medicine.
6. Contraindications to MRI (such as claustrophobia, metallic implant, etc.) based on MRI Screening
7. Participation in other interventional clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
8. Any physical or psychological symptom, based on the clinical judgment of the study physician that would make a participant unsuitable for the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women (<14 weeks gestation)
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Uteroplacental blood flow as assessed by doppler ultrasound, two dimensional phase contrast magnetic resonance imaging, and four dimensional flow magnetic resonance imaging. | Through study completion, an average of 4 years
  The goal of this research is to develop an arsenal of advanced U/S and MRI techniques that are compatible to be run simultaneously or sequentially to probe uteroplacental health and overcome the limitations posed by obesity and motion.The ideal combination of imaging procedures will help to progress with further human studies that actually benefit clinical diagnosis.

SECONDARY OUTCOMES:
Magnetic resonance perfusion and oxygenation as assessed by various U/S and MRI imaging techniques. | Through study completion, an average of 4 years
  Correlation between reduction in uteroplacental flow and perfusion with Fetal Growth Restriction and Preeclampsia.. Are reductions in uteroplacental flow, perfusion, or Oxygenation at 14, 20, 24 weeks correlated to Fetal Growth Restriction/Preeclamptic (FGR/PE) outcome?
Ferumoxytol (FE) detection at the maternal fetal interface as assessed by R2* and QSM | Through study completion, an average of 4 years
  Determination of immune cell redistribution at the Maternal Fetal Interface (MFI) via Fe-MR as a predictor of adverse pregnancy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Shah, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UnityPoint Health-Meriter Hospital, Madison, Wisconsin
  - University of Wisconsin-Hospitals and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT02791568/ICF_000.pdf